CLINICAL TRIAL: NCT02856373
Title: Renal Nerve Stimulation and Renal Denervation in Patients With Sympathetic Ventricular Arrhythmias: an Investigator Initiated Trial
Brief Title: Renal Nerve Stimulation and Renal Denervation in Patients With Sympathetic Ventricular Arrhythmias
Acronym: Redress VT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low enrollment number
Sponsor: Diagram B.V. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9218
Record Dates: First submitted 2016-06-10; First posted 2016-08-04 (Estimated); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Arrhythmias, Cardiac
Keywords: Denervation; Renal Artery
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- CPVT (Other): catecholaminergic polymorphic ventricular tachycardia (CPVT) patients
  Interventions: Procedure: RNS and RDN
- long QT syndrome (Other): long QT syndrome patients
  Interventions: Procedure: RNS and RDN
- ARVC (Other): arrhythmogenic right ventricular cardiomyopathy (ARVC) patients
  Interventions: Procedure: RNS and RDN
- HCM (Other): hypertrophic cardiomyopathy (HCM) patients
  Interventions: Procedure: RNS and RDN
- DCM (Other): dilated non-ischemic cardiomyopathy (DCM) patients
  Interventions: Procedure: RNS and RDN
- ICM (Other): ischemic cardiomyopathy (ICM) patients
  Interventions: Procedure: RNS and RDN

INTERVENTIONS:
Procedure: RNS and RDN — The patients will undergo electrical renal nerve stimulation and subsequently renal nerve denervation

SUMMARY:
Rationale:

Sympathetic activity plays an important role in the pathogenesis of ventricular tachyarrhythmia. Previous studies have shown evidence of significant heritable influences on individual responses to adrenergic stimulation. Catheter-based renal sympathetic denervation (RDN) is a novel treatment option for patients with resistant hypertension, proved to reduce local and whole-body sympathetic activity. The investigators hypothesize that percutaneous transluminal electrical stimulation of the sympathetic nerve bundles in the renal arteries will cause ventricular arrhythmias and renal denervation will suppress these arrhythmias in patients with sympathetic ventricular arrhythmias.

Objective:

This study will investigate the effects of renal nerve stimulation before and after percutaneous transluminal RDN on cardiac excitable properties including induction of ventricular tachy-arrhythmias before and after RDN in six studies, i.e. patients with catecholaminergic polymorphic ventricular tachycardia (CPVT), long QT syndrome and arrhythmogenic right ventricular cardiomyopathy (ARVC), sympathetically driven ventricular arrhythmias, hypertrophic cardiomyopathy (HCM), dilated non-ischemic cardiomyopathy (DCM) and ischemic cardiomyopathy (ICM). The aim of the six studies is to assess the anti-arrhythmic effects of RDN in patients with sympathetic ventricular tachy-arrhythmias.

Study design:

Investigator initiated, multi centre, six pretest-posttest design studies.

Study population:

Patients with recurrent sympathetically driven ventricular arrhythmia despite optimal pharmacological therapy. Patients should be diagnosed with CPVT and certain types of long QT syndrome, ARVC, HCM, DCM and ICM. Eligible patients will be in the age category of 18-85 year.

Intervention:

RDN will be performed according to routine clinical practice. Prior to the ablation procedure, catheter mapping of the renal arteries will be performed according to routine clinical practice. Clinical and biological responses to transluminal electrical renal nerve stimulation will be assessed before and after RDN.

Study endpoints:

* Main procedural study endpoint: Induction of ventricular arrhythmias in response to renal nerve stimulation prior to RDN and absence of renal nerves stimulation induced ventricular arrhythmias after RDN.
* Main clinical study endpoint: Development of ventricular arrhythmia during exercise stress testing performed 6 months after procedure.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

In several studies, it was shown that RDN was safe. The intervention resulted in significantly better control of blood pressure with less medication, and beneficial changes in heart rate variability, autonomic sympathetic balance, renal arteriolar function, and a higher success of atrial fibrillation prevention. In case reports and case series, RDN had a favourable effect in patients with sympathetic drug refractory ventricular tachy-arrhythmias.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is willing and able to comply with the protocol and has provided written informed consent.
2. The patient falls within the target group as stated in 4.1.
3. Patient is an acceptable candidate for RDN treatment
4. Patient is 18-85 years of age
5. Documentation of ventricular arrhythmia (ECG, rhythm strip or ICD interrogation)

Exclusion Criteria:

1. Contraindication to anticoagulation therapy or heparin.
2. Previous selective cardiac sympathetic denervation or previous RDN procedure.
3. Acute coronary syndrome, cardiac surgery, PCI or stroke within 3 months prior to enrolment.
4. Untreated hypothyroidism or hyperthyroidism.
5. More than grade 1/3 valvular regurgitation and/or significant valve stenosis (moderate or severe).
6. Severe LV dysfunction (LVEF <20% and/or grade 3/4 diastolic dysfunction).
7. Enrolment in another investigational drug or device study.
8. Woman currently pregnant or breastfeeding or not using reliable contraceptive measures during fertile age.
9. Mental or physical inability to participate in the study.
10. Planned cardiovascular intervention.
11. Life expectancy ≤ 12 months.
12. Renal artery stenosis >50% of the arterial lumen, or renal artery lumen ≤3 mm.
13. Complex renal artery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-03-03 (Actual); Primary Completion 2020-05-04 (Actual); Study Completion 2020-05-04 (Actual)

PRIMARY OUTCOMES:
Induction of ventricular arrhythmias (e.g. ventricular tachycardia and ventricular fibrillation) | A few minutes before RDN RNS will be performed. Time frame before RDN: 0-10 min. after RNS and before RDN. Time frame after RDN: 0-10 min.
  Induction of ventricular arrhythmias in response to RNS prior to RDN and absence of RNS induced ventricular arrhythmias after RDN
Development of ventricular arrhythmia | 6 months after procedure/intervention
  Development of ventricular arrhythmia during exercise stress testing performed 6 months after procedure/intervention

SECONDARY OUTCOMES:
Time to first detection of ventricular arrhythmia or appropriate ICD therapy | procedure/intervention-12 month follow up
  Time to first detection of ventricular arrhythmia or appropriate ICD therapy with the monitoring period starting immediately after the intervention.
Changes in ventricular refractoriness (frequency) | procedure/intervention
  Changes in ventricular refractoriness (frequency, beats/min) to programmed electrical stimulation in the setting of routine electrophysiological study before and directly (0-10 min) after RDN.
Changes in ventricular refractoriness (duration) | procedure/intervention
  Changes in ventricular refractoriness (duration, sec) to programmed electrical stimulation in the setting of routine electrophysiological study before and directly (0-10 min) after RDN.
Number of ventricular arrhythmias | procedure/intervention
  Inducibility (number) of ventricular arrhythmias to programmed electrical stimulation in the setting of routine electrophysiological study before and after RDN.
Ventricular arrhythmia burden | procedure/intervention- 6,12 months follow up
  Ventricular arrhythmia burden after 6 and 12 months of follow-up in patients with ICD or continuous rhythm monitoring with a loop recorder. The monitoring period starts immediately after the intervention.
Blood pressure | 6-12 months follow up
  Blood pressure at 6 and 12 months after the intervention
Number of (Supra-)Ventricular arrhythmias induced by exercise testing | baseline- 6 months follow up
  Number of (Supra-)Ventricular arrhythmias induced by exercise testing
(Supra-)Ventricular arrhythmias response changes (frequency) induced by exercise testing | baseline- 6 months follow up
  (Supra-)Ventricular arrhythmias response changes (frequency, beats/min) induced by exercise testing
(Supra-)Ventricular arrhythmias response changes (duration) induced by exercise testing | baseline- 6 months follow up
  (Supra-)Ventricular arrhythmias response changes (duration, sec) induced by exercise testing
Changes in heart rate variability | baseline- 3, 6 and 12 month follow up
  Changes in heart rate variability measures tested by Holter monitoring compared to measurement before the intervention
Changes in prevalence of events | 12 month before procedure/intervention-12 month follow up
  Changes in prevalence of events (hospital admission for VT or appropriate ICDshock) in the period of one year after intervention compared to a one year period before intervention.
Change in blood pressure | baseline- 6, 12 month follow up
  Change in blood pressure compared to measurement before the intervention
Heart rate response changes induced by exercise testing | baseline- 6 months follow up
  Heart rate response changes induced by exercise testing
Blood pressure response changes induced by exercise testing | baseline-6 months follow up
  Blood pressure response changes induced by exercise testing

CONTACTS AND LOCATIONS:
Overall Officials: Arif Elvan, MD, PhD, Principal Investigator — Isala, department of Cardiology
Locations (1):
- A. Elvan, Zwolle, Overijssel, Netherlands

IPD SHARING:
Plan to Share IPD: No